CLINICAL TRIAL: NCT04905745
Title: The Effectiveness and Safety of Integrative Korean Medicine Treatment for Bell's Palsy : A Prospective Observational Preliminary Study
Brief Title: The Effectiveness and Safety of Integrative Korean Medicine Treatment for Bell's Palsy
Status: Recruiting | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director of Jaseng Spine and Joint Research Institute, Jaseng Medical Foundation
Other Study IDs: JS-CT-2021-05
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Facial Paralysis, Peripheral
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Facial palsy: Adulthood facial palsy patients group who receive Korean integrative medicine.
  Interventions: Procedure: Korean integrative medicine

INTERVENTIONS:
Procedure: Korean integrative medicine — Any kind of Korean integrative medicine will be applicable and the treatment will be entirely determined by experienced clinicians. On the premise of the above, the following examples are the treatments applicable to the subject of this observational study.
  * Chuna: Chuna therapy is performed on the face and cervical spine to induce decompression of the captured facial nerve. In addition, SJS Non-Resistance Technique-Facial palsy (SJS NRT-F), a technique of Chuna, can be performed to stimulate the intrinsic receptive sensation of the facial muscles to promote the neuromuscular response.
  * Acupuncture: acupuncture can be applied on paralyzed muscle and others to improve symptoms and paralysis status.
  * Pharmacopuncture: pharmacopuncture can be applied on paralyzed muscle and others to improve symptoms and paralysis status.
  * Herbal medicine: It is prescribed according to clinical judgment according to the patient's symptoms and disease status.

SUMMARY:
This is an observational study that evaluate the effectiveness and safety of Korean integrative treatments in patients with peripheral facial nerve palsy. Adulthood patients aged between 19 to 69 who were diagnosed with peripheral facial nerve palsy and receive Korean integrative treatments for facial palsy will be enrolled in the study and the change will be followed according to the Facial disability index (FDI) at the 3 month moment after baseline.

DETAILED DESCRIPTION:
This is an observational study that evaluate the effectiveness and safety of Korean integrative treatments in patients with peripheral facial nerve palsy. A total of 100 patients who are in age of from 19 to 69, diagnosed with peripheral facial nerve palsy, in acute to subacute stage, and who receive Korean integrative treatments for facial palsy will be enrolled in this study. This study is an observational study and the intervention will be decided not by researchers, but by physicians in the real clinical practice. The treatment will be entirely determined according to each subject's medical conditions by an experienced clinician who has received more than 6 years of education and more than 3 years of training. This study will only record the contents of the intervention. Among all the data generated during the study period, data deemed necessary can be collected in the case record forms. The intervention will also be determined by the clinician, and the researcher presented assessment and data collection timepoints, which is independent of the treatment schedule. The on-treatment visit schedule will be once a week during the treatment is ongoing, and follow-up visit schedule will be on the 5th, 14th, and 53rd weeks after the baseline.

ELIGIBILITY:
Inclusion Criteria:

1. age of 19 to 69
2. diagnosed with unilateral peripheral facial nerve palsy
3. onset of facial palsy within 3 weeks or less.
4. an individual who can provide written consent form to participate in the study.

Exclusion Criteria:

1. diagnosed with central nervous system disease causing facial palsy
2. secondary facial palsy after multiple sclerosis, tumor, cerebrovascular disease and temporal bone fracture.
3. Ramsay-Hunt syndrome
4. bilateral or recurrent facial nerve palsy.
5. an individual who received any treatment that can have a significant effect on changes in facial paralysis within recent 2 month. (ie. facial nerve decompression surgery)
6. already or planned to be pregnant or breast-feeding within the study period.
7. uncontrolled diabetes mellitus within the last 3 months.
8. within a month after participating any other facial palsy-related clinical trials, or planning to participate other clinical trials within 6 month.
9. impossible to read and understand the documents, regarding informed consent form and the questionnaires.
10. difficult to participate according to the judgement of researchers.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adulthood male and female patients with peripheral facial nerve palsy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Facial disability index | week 14
  This is a questionnaire made to evaluate the subjective sensations of patients on the ability to use facial muscles and their emotional state. It is composed of 10 items, and 1-5 is composed of 5 points per item for movement state, and 6-10 is composed of 6 points per item for sociological state and emotional state.

SECONDARY OUTCOMES:
Facial disability index (FDI) | week 1, 5, 14, 53
  This is a questionnaire made to evaluate the subjective sensations of patients on the ability to use facial muscles and their emotional state. It is composed of 10 items, and 1-5 is composed of 5 points per item for movement state, and 6-10 is composed of 6 points per item for sociological state and emotional state.
House-Brackmann facial palsy grade system (HB grade) | week 1, 5, 14, 53 and every week during treatment (for survival analysis in complete recovery)
  HB grade is a scale to evaluate facial palsy into 6 stages based on the severity of facial palsy, especially the muscles around the mouth and the muscles arount the eyes.
Numeric rating scale (NRS) | week 1, 5, 14, 53 and every week during treatment
  NRS is a 11-point scale of 0-10. the researcher will rate NRS for postauricular pain and discomforts in the face and cervical area.
Facial nerve grading system (FNGS 2.0) | week 1, 5, 14, 53
  FNGS 2.0 is calculated based on the total score by section by section in facial part and additional score with synkinesis movement. The result of FNGS 2.0 well indicate the palsy status, with the grade of 1-6 and 4-24 points.
Synkinesis Assessment Questionnaire (SAQ) | week 1, 5, 14, 53
  The SAQ is a questionnaire that calculates the total score of 9 representative symptoms of synkinesis into 1-5 points for each item.
Patient Global Impression of Change (PGIC) | week 5, 14, 53
  Patient global impression of change (PGIC) is a method that allows the patient to subjectively evaluate the degree of improvement in 7 degree of scale.
Short Form-12 Health Survey (SF-12) | week 1, 5, 14, 53
  The SF-12 is a questionnaire that evaluates the overall health-related quality of lives (HRQoL). SF-12 consists of 12 questions covering following 8 areas, to evaluate functional health and well-being of individuals both ill and healthy; physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, KMD,Ph.D, Study Director — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No